CLINICAL TRIAL: NCT04795284
Title: Biomechanical Parameters of Gait in Patients with Symptomatic Lumbar Spinal Stenosis and Healthy Elderly.
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR_gaitup_2020
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Spinal Stenosis; Healthy Elderly
Keywords: Lumbar Spinal Stenosis; Healthy elderly; Walking capacity; Biomechanical parameters
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with symptomatic lumbar spinal stenosis: 30-meter walking task (15 meters round trip) following by a rest period of 2 minutes. Participants are invited to perform the 30-meter walking task twice. Inertial sensors are put on each participant foot.
- Healthy elderly: 30-meter walking task (15 meters round trip) following by a rest period of 2 minutes. Participants are invited to perform the 30-meter walking task twice. Inertial sensors are put on each participant foot.

SUMMARY:
The aim of this study is to compare biomechanical walking parameters between patients with symptomatic lumbar spinal stenosis and healthy elderly.

ELIGIBILITY:
Inclusion Criteria:

Patients with lumbar spinal stenosis

* Having a diagnosis of lumbar spinal stenosis (at least 1 level)
* Having neurologic claudication due to the lumbar spinal stenosis

Healthy elderly

* Being over 50 years old of age
* No back or leg pain during walking

Exclusion Criteria:

* Symptomatic hip or knee Ostearthritis
* Not able to give their free consent
* Being in a wheelchair (not able to walk 30 meters)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with a symptomatic lumbar spinal stenosis Group 2: Healthy elderly from the community
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
biomechanical walking parameters (gait cycle, stride length, walking time, walking speed, swing width, minimal toe clearance) | During the 30-meter walking test
  Gait cycle = % stance phase, % swing phase / Stride length = describes the distance between two successive footprints on the ground / walking time = time to complete the 30-meters walking test in seconds / walking speed = walking stride velocity measured in meter/second / swing width = the maximal lateral excursion of the foot during the swing phase / minimal toe clearance = minimum height of the toes during the swing phase (in meter)
Quality of life (Euro-Qol - 5D) | One time (before the completion of the 30-meter walking test)
  Quality of life related to mobility, self-care, usual activities, pain and discomfort, anxiety and depression. Each category has a score ranging from 1 to 3 and higher values indicate a worst outcome.
International Physical Activity Questionnaire (IPAQ) | One time (before the completion of the 30-meter walking test)
  Physical activity habits. IPAQ score range from 1 to 3 where a score of 3 indicates a higher practice of physical activity

SECONDARY OUTCOMES:
French-Canadian adaptation of Swiss Spinal Stenosis Questionnaires (FC-SSSQ) | One time (before the completion of the 30-meter walking test) - Only for patients with lumbar spinal stenosis
  Pain, function and satisfaction related to lumbar spinal stenosis. Pain subscale score range from 7 to 35 with higher values indicate a worst outcome, Function subscale score range from 5 to 20 with higher values indicate a worst outcome, Satisfaction subscale score range from 6 to 24 with higher values indicate a worst outcome. The total score is composed of the three subscales and range from 18 to 79.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No